CLINICAL TRIAL: NCT02788084
Title: Development of a Tissue-Based & Cell Free DNA Next-Generation Sequencing Workflow
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alberta Health Services, Calgary (Other)
Responsible Party: Principal Investigator, Gwynivere Davies, Resident, Alberta Health Services, Calgary
Other Study IDs: CC-16-0582
Record Dates: First submitted 2016-05-25; First posted 2016-06-02 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Next Generation Sequencing; Cell free DNA
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA library, RNA and formalin fixed paraffin embedded (FFPE) specimens will be banked with participants' prior permission.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- B cell Non-Hodgkin Lymphoma: 18 years of age or older with new diagnosis of non-Hodgkin lymphoma with FFPE specimen demonstrating enough tissue for elucidation of lymphoma specific variant and immunoglobulin clonotype, willing to provide baseline and follow up bloodwork to look for presence of variant and clonotype.

SUMMARY:
1. Develop a Next-Generation Sequencing (NGS) workflow for mutation profiling of formalin-fixed paraffin-embedded (FFPE) tissue and cell-free DNA (cfDNA) specimens.
2. Calculate the proportion of cases in a test series of B-cell non-Hodgkin Lymphomas (BNHL) with somatic mutations or immunoglobulin heavy chain (IGH) gene rearrangements common to both FPPE and cfDNA specimens.
3. Determine if certain types of BNHL are more likely to have mutation profiles common to both FFPE & corresponding cfDNA ("FFPE-cfDNA dyads")
4. Determine if specific mutations or mutation profiles in FFPE or cfDNA specimens (or both) are of prognostic value after a clinical follow-up of 2 years from the time of diagnosis.

DETAILED DESCRIPTION:
Patients with newly diagnosed B cell NHL will be identified. Samples will be cored from their diagnostic FFPE blocks and assayed to find lymphoma specific variants and immunoglobulin heavy chain gene rearrangements. Blood samples collected at baseline will be compared to see if variants and rearrangements can be detected in tumor specific DNA based on previous studies. Participant data will be collected, and clinical outcomes will be assessed to determine effect of mutation profiles on outcomes over 2 year follow up.

Blood samples will be prospectively collected at scheduled follow up and if primary objectives of this study are met, will be assessed for presence of cfDNA and impact of variation on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of B cell NHL
* Willing to have blood collected at timepoints of regularly scheduled follow up
* Formalin fixed paraffin embedded (FFPE) diagnostic specimen sufficient for further testing

Exclusion Criteria:

* Unwilling or unable to participate in follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years or older with new diagnosis of B cell non Hodgkin lymphoma (NHL) with follow up occurring in Calgary undergoing chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
2 year Progression Free Survival | 2 years from diagnosis of B cell non-Hodgkin Lymphoma
  Recorded in percentage. To determine impact of lymphoma specific mutation on outcome.
2 year Overall Survival | 2 years from diagnosis of B cell non-Hodgkin Lymphoma
  Recorded in percentage. To determine impact of lymphoma specific mutation on outcome.
Occurrence of lymphoma specific mutations or detectable IgH rearrangements in circulating tumor specific DNA in blood samples at baseline | Determined at baseline
  Proportion of cases of BNHL with somatic mutations or IgH gene rearrangements detectable in blood. Will be recorded in percentage, and determined at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Mahe, MD, FRCPC, Principal Investigator — Calgary Laboratory Services, University of Calgary
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No